CLINICAL TRIAL: NCT07141602
Title: Correlation Between Stages of Mandibular Second Molar Calcification and Cervical Vertebrae Maturation Index for Assessment of Skeletal Maturation: A Cross Sectional Study
Brief Title: Correlation Between Stages of Mandibular 2nd Molar Calcification and CVMI for Assessment of Skeletal Maturation: A Cross Sectional Study
Status: Active, not recruiting | Type: Observational
Sponsor: Mohamed Abd El-Ghafour (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abd El-Ghafour, Mohamed Abd El-Ghafour Omar, BDS, MSc, PhD, Cairo University
Organization: Cairo University (Other)
Other Study IDs: ORTH7-3-2
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Correlation Between Second Molar Calcification Stage and CVMI for Skeletal Maturation Assessment in Egyptian Population
Keywords: second molar tooth, cervical vertebrae maturation, skeletal maturation, lateral cephalogram, panorama

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- will include males
  Interventions: Diagnostic Test: lateral cephalometric x- ray and dental panoramic tomogram
- will include females
  Interventions: Diagnostic Test: lateral cephalometric x- ray and dental panoramic tomogram

INTERVENTIONS:
Diagnostic Test: lateral cephalometric x- ray and dental panoramic tomogram — lateral cephalometric x- ray and dental panoramic tomogram

SUMMARY:
The aims of this study will be:

1. To investigate the relationships between mandibular second molar calcification stages and skeletal maturity in Egyptian population, and
2. To evaluate whether the mandibular second molar calcification stages can be used as a reliable diagnostic tool to assess skeletal maturity in Egyptian population.

DETAILED DESCRIPTION:
This cross-sectional study will include 106 Egyptian subjects with age range between 9 and 18 years old, who will present to outpatient clinic of Orthodontic department, Faculty of Dentistry, Cairo University, and will be classified according to their gender into two groups (males and females). Radiographs (panorama and cephalogram) will be collected from all study participants who meet inclusion criteria for data analysis. The inclusion criteria will be as follows:

* Chronological age ranging from 9 to 18 years
* No serious illness
* Normal overall growth and development
* Absence of abnormal dental conditions, such as impaction, transposition, and congenitally missing teeth
* Absence of previous history of trauma or disease to the face and neck
* Absence of orthodontic treatment
* No permanent teeth extracted

We will obtain panoramic and lateral cephalometric radiographs of 106 Egyptian subjects from the pretreatment records of patients attending clinics for orthodontic treatment.

All radiographic assessments will be performed in a darkened room. Any radiograph that shows motion dullness or has poor contrast will be discarded. A single radiologist will expose and develop all radiographs.

ELIGIBILITY:
Inclusion Criteria:

* • Chronological age ranging from 9 to 18 years

  * No serious illness
  * Normal overall growth and development
  * Absence of abnormal dental conditions, such as impaction, transposition, and congenitally missing teeth
  * Absence of previous history of trauma or disease to the face and neck
  * Absence of orthodontic treatment
  * No permanent teeth extracted

Exclusion Criteria:

-

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: 212 Egyptian subjects with their age ranging between 9 and 18 years old, who will present to outpatient clinic of Orthodontic department, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
to evaluate the frequency of stage E of dental index in female subjects. | one year
  to evaluate the frequency of stage E of dental index in female subjects.

SECONDARY OUTCOMES:
to evaluate relationships between the stages of calcification of mandibular second molar (DI) and cervical vertebrae maturation index (CVMI). | one year
  to evaluate relationships between the stages of calcification of mandibular second molar (DI) and cervical vertebrae maturation index (CVMI).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry-Cairo University, Gizah-Egypt, Egypt